CLINICAL TRIAL: NCT06512246
Title: Failure Factors of Endoscopic Retrograde Cholangiopancreatography After Gastrointestinal Reconstruction and Effectiveness of Remedial Measures
Brief Title: Failure Factors of ERCP After Gastrointestinal Reconstruction and Effectiveness Analysis of Remedial Measures
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BFHHZS20240136
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: Endoscopic Retrograde Cholangiopancreatography; Gastrointestinal Reconstruction; Remedial Measure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study, including 195 patients with gastrointestinal reconstruction, who treated with Endoscopic Retrograde Cholangiopancreatography (ERCP) at Beijing friendship hospital. The investigators assessed the outcomes of failure factors of ERCP and effectiveness of remedial measures.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is an invasive procedure in which an endoscope is inserted into the descending part of the duodenum through the duodenal papilla, and special instruments are used to enter the bile duct or pancreatic duct for examination and treatment with the assistance of X-ray.

For normal upper digestive tract anatomy, the technical success rate of ERCP was 97.6% and the treatment success rate was 95.2%. But when the upper GI tract anatomy is altered due to surgery, standard ERCP is operationally challenging and sometimes impossible. For the treatment of gastroduodenal malignant tumors, obesity and peptic ulcer, subtotal gastrectomy and total gastrectomy are often used in combination with gastrointestinal reconstruction. The most common gastrointestinal reconstruction procedures include Billroth I, Billroth II, Roux-en-Y and so on. Billroth I is a gastroduodenal anastomosis, which is more consistent with the original physiological condition of the gastrointestinal tract, and usually does not increase the difficulty of ERCP operation. Billroth II closed the duodenal end and anastomosed the stomach and jejunum to form an input loop and an output loop behind the gastrointestinal anastomosis. Roux-en-Y is to close the duodenal end and transect the jejunum with Treitz ligament at a distance of 10-15cm. The distal end is anastomosed with the remnant stomach, and the proximal end is anastomosed with the jejunum at a distance of 45-60cm from the gastrointestinal anastomosis. Due to the change of gastrointestinal structure after gastrointestinal reconstruction, patients may be complicated with cholelithiasis, pancreaticobile duct stenosis and other diseases, requiring ERCP to assist in diagnosis and treatment. However, the alteration of digestive tract anatomical structure and possible postoperative complications, including anastomotic fistula and anastomotic stenosis, may lead to certain difficulty in ERCP operation. The success of ERCP includes the success of ERCP implantation, ERCP intubation and ERCP treatment. According to previous studies at home and abroad, the relevant success rates of ERCP after gastrointestinal reconstruction are 82.3%-90.5%, 77.5%-88.6% and 46.3%-88.6%, respectively. Current studies suggest that the gastrointestinal remodeling procedure, the type of operating endoscope, and the experience of operating physicians are related to the success rate of ERCP operation. When ERCP fails, it can be treated with ERCP again, percutaneous hepatic puncture biliary drainage (PTCD), endoscopic ultrasound, and surgery.

In a retrospective analysis, 195 patients with gastrointestinal reconstruction, who treated with Endoscopic Retrograde Cholangiopancreatography (ERCP) at Beijing Friendship Hospital were studied. The investigators assessed the outcomes of failure factors of ERCP and effectiveness of remedial measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* After gastrointestinal reconstruction (Billroth Ⅱ Anastomosis, Roux-en-Y Anastomosis).
* Endoscopic retrograde cholangiopancreatography (ERCP) was performed for common bile duct stone with choledocholithiasis, pancreatic duct stenosis, or obstructive jaundice with endoscopic indication.

Exclusion Criteria:

* After Billroth I Anastomosis.
* Accompanied by serious cardiopulmonary disease or coagulation dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with gastrointestinal reconstruction underwent ERCP at Beijing Friendship Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of Reaching Duodenal Papilla | during the operation
  successfully reaching duodenal papilla during the endoscopic procedure

SECONDARY OUTCOMES:
Successful Intubation Rate | during the operation
  successful intubation during the ERCP procedure
Successful Endoscopic Treatment Rate | during the operation
  successful endoscopic treatment during the ERCP procedure
Effective Rate of Remedial Measures | during the operation
  remedial measures successfully relief symptom
ERCP-related complication rate | during the operation
  The complications include pancreatitis, hemorrhage, perforation, pneumonia, etc. The results of intraoperative endoscopic observation, postoperative symptoms and signs, blood routine examination, amylase, lipase, and imaging and endoscopic examination were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fujing Lv, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China